CLINICAL TRIAL: NCT02454478
Title: Phase 1 Study of Lenvatinib in Combination With Everolimus in Subjects With Unresectable Advanced or Metastatic RCC
Brief Title: Study of Lenvatinib in Combination With Everolimus in Participants With Unresectable Advanced or Metastatic Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-112
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: lenvatinib; Everolimus; Carcinoma; Unresectable advanced renal cell carcinoma; Metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma | interventions — lenvatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib plus Everolimus (Experimental)
  Interventions: Drug: Lenvatinib; Drug: Everolimus

INTERVENTIONS:
Drug: Lenvatinib
Drug: Everolimus
  Other Names: Lenvatinib plus Everolimus orally once a day

SUMMARY:
Phase 1 study to investigate the tolerability and safety of lenvatinib in combination with Everolimus in participants with unresectable advanced or metastatic RCC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent of this study.
2. Willing and able to comply with all aspects of the protocol after being fully informed of the content.
3. Males or females aged greater than or equal to 20 years at the time of informed consent.
4. Histological or cytological confirmation of RCC.
5. Participants must have confirmed diagnosis of unresectable advanced and/or metastatic RCC.
6. Disease progression following vascular endothelial growth factor (VEGF) targeted therapy.
7. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) of 0 to 1.
8. Adequately controlled blood pressure with or without the use of antihypertensive agents.
9. Participants with adequate function of major organs.
10. Adequate blood coagulation function, defined as international normalized ratio (INR) less than or equal to 1.5.
11. Survival expectation of 3 months or longer after study enrollment.
12. Participants with adequate washout period from the end of prior treatment to the start of study drug administration.
13. Females of childbearing potential must not have had unprotected sexual intercourse within 28 days before participant registration and must agree to use a highly effective method of contraception throughout the entire study period and for 30 days after final administration of investigational drug. If currently abstinent, the participant must agree to use a double-barrier method as described above if she becomes sexually active during this study period or for 30 days after investigational drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before administration and must continue to use the same contraceptive during this study and for 30 days after investigational drug discontinuation.
14. Male participants and their female partners must meet the criteria above.

Exclusion Criteria:

1. Participants with central nervous system (CNS) metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example, radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
2. Prior exposure to lenvatinib.
3. Participants who have not recovered from toxicities to less than or equal to Grade 1 as a result of prior anticancer therapy, except alopecia.
4. Major surgery within 3 weeks prior to the first dose of lenvatinib.
5. Participants with a urine protein greater than or equal to 1 gram per 24 hours (g/24 hours).
6. Uncontrollable diabetes as defined by fasting glucose greater than 1.5* upper limit of normal (ULN).
7. Fasting total cholesterol greater than 7.75 millimole per liter (mmol/L) (greater than 300 milligram per decilitre [mg/dL]).
8. Fasting triglycerides greater than 2.5 * ULN.
9. Any condition that might affect the absorption of lenvatinib and/or everolimus.
10. Significant cardiovascular impairment.
11. Bleeding or thrombotic disorders or use of anticoagulants requiring therapeutic INR monitoring.
12. Active hemoptysis.
13. Active infections that require systemic treatment.
14. Human immunodeficiency virus (HIV) positive.
15. Hepatitis B virus (HBV).
16. A history of interstitial pneumonia with clinical manifestation or as confirmed by means of diagnostic imaging.
17. Medical need for the continued use of potent or moderate inhibitors of cytochrome P450 3A (CYP3A) or P-gp, or potent or moderate inducer of CYP3A.
18. Known intolerance to lenvatinib (or any of the excipients) or known hypersensitivity to everolimus (or any of the excipients) or rapmycins (sirolimus, temsirolimus and so on).
19. Alcohol or drug dependency or abuse, inability to comply with every aspects of the study protocol, or any physical or mental conditions that in the opinion of the investigators would preclude the participant's participation in the study.
20. Females who are pregnant or breastfeeding (not eligible even she discontinues breastfeeding).
21. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Eisai Trial Site #1, Chiba
  - Eisai Trial Site #1, Tokyo
  - Eisai Trial Site #2, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 sites in Japan from 01 July 2015 to 29 May 2017.
Pre-assignment Details: A total of 9 participants were screened, of which 7 were enrolled and treated in the study.
Groups:
- Lenvatinib 18 mg + Everolimus 5 mg: Participants received lenvatinib 18 milligram (mg) capsules along with everolimus 5 mg tablets, orally, once daily in 28-days treatment cycles up to disease progression, development of unacceptable toxicity, participant's request to discontinue, withdrawal of consent, or study termination by sponsor (up to 23 cycles).
Period: Overall Study
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Started | 7
Completed | 6
Not Completed | 1
Not completed — Incomplete DLT Evaluation | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who received at least 1 dose of lenvatinib.
Groups:
- Lenvatinib 18 mg + Everolimus 5 mg: Participants received lenvatinib 18 mg capsules along with everolimus 5 mg tablets, orally, once daily in 28-days treatment cycles up to disease progression, development of unacceptable toxicity, participant's request to discontinue, withdrawal of consent, or study termination by sponsor (up to 23 cycles).
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (6.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Any Dose Limiting Toxicity (DLT)
Description: DLT was defined as toxicity related to the combination therapy and was graded according to Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03).
Time Frame: From first dose of study drug up to Cycle 1 Day 28 (Cycle length=28 days)
Population: The DLT analysis set was the group of participants who had completed treatment Cycle 1 without major protocol deviation with a treatment compliance of at least 75 percent (%) and had been assessed for DLT, and participants who had experienced DLT during Cycle 1.
Measure: Number; unit: participants
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 6
participants | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug (up to approximately 21.5 months)
Population: The safety analysis set was the group of participants who received at least 1 dose of lenvatinib.
Measure: Number; unit: participants
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
participants
  TEAE | 7
  SAE | 3

3. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Levatinib and Everolimus
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 4 ,8, and 24 hours postdose (Cycle length=28 days)
Population: The pharmacokinetic (PK) analysis was group of participants who received at least 1 dose of lenvatinib and had sufficient data from which at least one PK parameter could be calculated.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
nanogram per milliliter (ng/mL)
  Lenvatinib: Cycle 1 Day 1 | 289 (136)
  Everolimus: Cycle 1 Day 1 | 39.1 (18.7)

4. Secondary Outcome: Css,Max: Maximum Observed Plasma Concentration at Steady State for Levatinib and Everolimus
Time Frame: Cycle 1 Day 15 predose and at 1, 2, 4 ,8, and 24 hours postdose (Cycle length=28 days)
Population: The PK analysis was group of participants who received at least 1 dose of lenvatinib and had sufficient data from which at least one PK parameter could be calculated. The PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
ng/mL
  Lenvatinib: Cycle 1 Day 15: number analyzed (Participants) | 5
  Lenvatinib: Cycle 1 Day 15 | 257 (112)
  Everolimus: Cycle 1 Day 15: number analyzed (Participants) | 5
  Everolimus: Cycle 1 Day 15 | 41.5 (19.3)

5. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Levatinib and Everolimus
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 4 ,8, and 24 hours postdose (Cycle length=28 days)
Population: The PK analysis was group of participants who received at least 1 dose of lenvatinib and had sufficient data from which at least one PK parameter could be calculated.
Measure: Median (Full Range); unit: hour
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
hour
  Lenvatinib: Cycle 1 Day 1 | 3.87 [0.95 to 3.87]
  Everolimus: Cycle 1 Day 1 | 0.92 [0.82 to 1.10]

6. Secondary Outcome: Tss,Max: Time to Reach the Maximum Plasma Concentration (Cmax) at Steady State for Levatinib and Everolimus
Time Frame: Cycle 1 Day 15 predose and at 1, 2, 4 ,8, and 24 hours postdose (Cycle length=28 days)
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
hour
  Lenvatinib: Cycle 1 Day 15: number analyzed (Participants) | 5
  Lenvatinib: Cycle 1 Day 15 | 3.77 [1.88 to 4.08]
  Everolimus: Cycle 1 Day 15: number analyzed (Participants) | 5
  Everolimus: Cycle 1 Day 15 | 0.97 [0.83 to 3.97]

7. Secondary Outcome: AUC 0-t: Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for Levatinib and Everolimus
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 predose and at 1, 2, 4 ,8, and 24 hours postdose (Cycle length=28 days)
Population: The PK analysis set was group of participants who received at least 1 dose of lenvatinib and had sufficient data from which at least one PK parameter could be calculated. The PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: hour * nanogram per milliliter (h*ng/mL)
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
hour * nanogram per milliliter (h*ng/mL)
  Lenvatinib: Cycle 1 Day 1 | 2770 (1090)
  Everolimus: Cycle 1 Day 1 | 211 (115)
  Lenvatinib: Cycle 1 Day 15: number analyzed (Participants) | 5
  Lenvatinib: Cycle 1 Day 15 | 3220 (1080)
  Everolimus: Cycle 1 Day 15: number analyzed (Participants) | 5
  Everolimus: Cycle 1 Day 15 | 401 (128)

8. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR included complete response (CR), partial response (PR), stable disease (SD), and PD (progressive disease). BOR was assessed using Response Evaluation Criteria in Solid Tumor (RECIST) 1.1
Time Frame: From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 23 months)
Population: The efficacy analysis set was the group of participants who received at least 1 dose of lenvatinib.
Measure: Number; unit: participants
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
participants
  CR | 0
  PR | 5
  SD | 1
  PD | 1

9. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved BOR of CR or PR. ORR was assessed using RECIST 1.1.
Time Frame: as for outcome 8
Population: The efficacy analysis set was the group of participants who received at least 1 dose of lenvatinib.
Measure: Number; unit: percentage of participants
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
percentage of participants | 71.4

10. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved BOR of CR, PR, or SD. DCR was assessed based on RECIST 1.1.
Time Frame: as for outcome 8
Population: The efficacy analysis set was the group of participants who received at least 1 dose of lenvatinib.
Measure: Number; unit: percentage of participants
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
percentage of participants | 85.7

11. Secondary Outcome: Number of Participants With the Minimum Percent Change From Baseline in the Sum of Diameters of Target Lesions
Time Frame: Baseline up to first tumor assessment at which diameter of target lesions were available (up to approximately 23 months)
Population: The efficacy analysis set was the group of participants who received at least 1 dose of lenvatinib.
Measure: Number; unit: participants
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
Number analyzed (Participants) | 7
participants
  Less than or equal to (<=) -30% | 5
  Greater than (>) -30% to less than (<) 20% | 1
  Greater than or equal to (>=) 20% | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug (up to approximately 21.5 months)
Groups:
- Lenvatinib 18 mg + Everolimus 5 mg: Participants received lenvatinib 18 mg capsules along with everolimus 5 mg tablets, orally, once daily in 28-days treatment cycles up to disease progression, development of unacceptable toxicity, participant's request to discontinue withdrawal of consent, or study termination by sponsor (up to 23 cycles).
Arm/Group | Lenvatinib 18 mg + Everolimus 5 mg
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 18 mg + Everolimus 5 mg (N=7)
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 18 mg + Everolimus 5 mg (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 5
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 4
Blood cholesterol increased (Investigations) | 5
Weight decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Lipase increased (Investigations) | 2
Amylase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Traumatic occlusion (Gastrointestinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Periodontitis (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 3
Eyelid oedema (Eye disorders) | 1
Wound (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT02454478/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02454478/SAP_001.pdf